CLINICAL TRIAL: NCT03030274
Title: Prospective, Non-randomized, Pilot Study to Assess Safety and Efficacy of a Novel Atrial Flow Regulator (AFR) in Heart Failure Patients With Reduced Ejection Fraction or in Heart Failure Patients With Preserved Ejection Fraction
Brief Title: The Prelieve Trial - Pilot Study to Assess Safety and Efficacy of a Novel Atrial Flow Regulator (AFR) in Heart Failure Patients
Acronym: PRELIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Occ2016_06
Record Dates: First submitted 2017-01-17; First posted 2017-01-24 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure Low Output; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occlutech AFR Device (Experimental): Prospective, non-randomized, pilot study to assess safety and efficacy of a novel Atrial Flow Regulator in Heart Failure Patients with with reduced Ejection Fraction (HFrEF) and Heart Failure Patients with preserved Ejection Fraction (HFpEF); the AFR-Prelieve Trial
  Interventions: Device: Occlutech AFR device

INTERVENTIONS:
Device: Occlutech AFR device — Catheter-guided placement of an AFR device following balloon atrial septostomy.

SUMMARY:
This study aims to investigate safety and efficacy of the Occlutech® AFR device in patients with HFrEF (Heart failure with reduced ejection fraction) and HFpEF (Heart failure with preserved ejection fraction)

DETAILED DESCRIPTION:
This study will enroll subjects with HFrEF or HFpEF, until a maximum of 100 patients have undergone implantation with the Occlutech® AFR device.

Enrolled patients will be stratified according to their ejection fraction as either HFrEF (ejection fraction > 15% and <40 %) or HFpEF ( ejection Fraktion > 40 % to 70 %). It is planned to enroll at least 100 patients per stratification subgroup.

ELIGIBILITY:
Inclusion criteria. Each patient must fulfill ALL of the following criteria and details:

1. Age ≥18 years
2. Heart failure resulting in NYHA class III or IV ambulatory
3. Ongoing management of heart failure according to ESC (European Society of Cardiology) (15) -guidelines during previous ≥6 months
4. Control with Arrhythmia with heart rate <110bpm
5. Life expectancy of at least 1 year
6. The patient should have the ability to fluently speak and understand the language in which the study is being conducted
7. Written, informed consent by the patient for participation in the study and agreement to comply with the follow-up schedule
8. Patient has had a successful Balloon Atrial Septostomy (BAS) procedure and is in a stable hemodynamic state, as assessed by the investigator
9. LVEF ≥15% and ≤ 70% , EF measured via Echocardiography 9.1.9.1. And for LVEF ≥ 40% (HFpEF): elevated NT-pro-BNP of ≥ 125 pg/ml
10. Elevated left ventricular filling pressure documented by 10.1. Either Pulmonary capillary wedge pressure (PCWP) or left ventricular end-diastolic pressure at rest ≥ 15 mmHg and greater then central venous preassure (CVP) 10.2. 10.2. Or: End-expiratory PCWP ≥25 mmHg at exercise and CVP <20 mm Hg
11. Transseptal catheterization and femoral vein access is determined to be feasible

Exclusion Criteria:

1. Local or generalized sepsis or other acute infection(s)
2. Any coagulation disorder, if clinically relevant in the opinion of the operator.
3. Allergy to nickel and/or titanium and/or nickel/titanium-based materials, if not medically manageable
4. Allergy to anti-platelet, -coagulant, or -thrombotic therapy, if not medically manageable
5. Intolerance to contrast agents, if not medically manageable
6. Participation in another medical trial testing a therapy less than 30 days before the intended AFR implantation procedure
7. Trans-oesophageal echocardiography and / or use of general anaesthetic is contraindicated
8. Breast feeding women
9. Pregnancy

   Processes which would technically disturb the safe intervention as planned:
10. Occluded inferior vena cava access
11. History of ASD and/or atrial septal repair or closure device in place
12. Intracardiac thrombus

    Clinical conditions:
13. Moderate valvular diseases requiring therapy according to current ESC guidelines. Patients are eligible in case therapy is formally indicated but cannot be performed due to technical or medial reasons if the latter is confirmed in writing by the PI in mutual agreement with the heart team and Severe aortic stenosis with valve area < 1.5cm² and Severe AR, TR or MR. Classification of severity of regurgitation should follow the definition provided in Lancelotti et al, Eur Heart J Cardiovasc Imaging 2013 [22]
14. Patients who has unstable and intractable angina pectoris
15. Evidence of right heart failure defined as (by ECHO)

    1. Severe Right Ventricular Dysfunction (TAPSE < 14 mm)
    2. Severe Right Ventricular Dilatation (RV volume ≥ LV volume)
    3. Severe pulmonary hypertension (PASP > 60 mm Hg)
16. Active malignancy
17. Severe valve disease, or implanted mechanical valve prosthesis
18. Congenital heart defect
19. Large PFO with significant atrial septal aneurysm (bubble test shows more than 20 bubbles)
20. Inability to perform 6-minutes walking test
21. Clinically relevant thrombocytopenia, thrombocytosis, leukopenia, or anemia
22. Symptomatic carotid artery disease
23. Mitral valve stenosis
24. Has any condition that, in the opinion of the Investigator, might interfere with the Implantation, might affect the patients well-being thereafter or might interfere with the conduct of the study
25. Systolic blood pressure of >170 mmHg, despite medical therapy
26. Severe lung disease (causing PHT with systolic PAP >60mmHg)
27. Pulmonary Hypertension (Systolic PAP >60mmHg)
28. TIA or stroke within the last 6 months
29. Scheduled for heart transplantation
30. Bleeding disorders (INR > 2.0, Thrombocytes < 100.000, Hemoglobin <8.0 gr/dl)
31. Myocardial infarction or percutaneous intervention or CABG (all within the last 3 month) or indication for a coronary intervention
32. Resyncronization therapy started within the last 6 months
33. Aneurysm of the septum
34. Hypertrophied Inter Atrial Septum (IAS) > 10mm depth
35. Hypertrophic Obstructive Cardiomyopathy (HOCM) or infiltrative CM as cause of HF
36. Thromboembolic events within the last 6 months
37. Dialysis and renal insufficiency requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Device Effects (SADE) within 3 month following implantation. | 0-3 month
  Incidence of Serious Adverse Device Effects (SADE) following implantation such as:
  * device dislocation / embolization
  * damage to the tricuspid or mitral valve caused by the device
  * intractable arrhythmias caused by the device
  * any circumstances that require device removal.

SECONDARY OUTCOMES:
Serious Adverse Device Effects (SADE) between 3-12 month following implantation | 3-12 month
  Incidence of all Serious Adverse Device Effects (SADE) following implantation
Device placement | 0-12 month
  Device placement in situ
Left to Right shunt through the AFR device | 0-12 month
  Evidence of Left to Right shunt through the AFR device

CONTACTS AND LOCATIONS:
Locations (26):
- Belgium (5):
  - AZ Maria Middelares, Ghent, Buitenring Sint-Denijs 30
  - UZ Leuven, Leuven, Herestraat 49
  - University Hospital Brussels, Brussels, Laarbeeklaan 101
  - Algemeen Stedelijk Ziekenhuis (Asz), Aalst, Merestraat 80
  - OLV (Onze-Lieve-Vrouwziekenhuis) Hospital Aalst, Aalst, Moorselbaan 164
- Germany (11):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Herzzentrum Uniklinik Köln, Cologne
  - CardioVasculäres Centrum Frankfurt, Frankfurt
  - Cardiologicum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University of Homburg, Homburg
  - Herzzentrum Leipzig, Leipzig
  - Uniklinikum Magdeburg A. ö. R., Magdeburg
  - Universitätsmedizin Rostock, Rostock
  - University of Würzburg, Würzburg
- Turkey (Türkiye) (10):
  - Dışkapı Yıldırım Beyazıt Eğitim ve Araştırma Hastanesi, Ankara, Altındağ
  - Hacettepe Üni Hastanesi, Ankara, Altındağ
  - Ege Üniversitesi Hastanesi, Izmir, Bornova
  - İstanbul Üniversitesi, Istanbul, Fatih
  - Kartal Koşuyolu Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Istanbul, Kartal
  - Tepecik Eğitim Ve Araştırma Hastanesi, Izmir, Konak
  - Sivas Cumhuriyet Üniversitesi Tıp Fakültesi Araştırma ve Uygulama Hastanesi, Sivas, Merkez
  - Bezmialem University, Istanbul
  - Kocaeli Üniversitesi Hastanesi, Kocaeli
  - İzmir Kâtip Çelebi Üniversitesi, Izmir, Çiğli

REFERENCES:
- [Derived] Lauder L, Bergmann MW, Paitazoglou C, Ozdemir R, Iliadis C, Bartunek J, Lauten A, Keller T, Weber S, Sievert H, Anker SD, Mahfoud F. Predicted impact of atrial flow regulator on survival in heart failure with reduced and preserved ejection fraction. ESC Heart Fail. 2023 Aug;10(4):2559-2566. doi: 10.1002/ehf2.14384. Epub 2023 Jun 13. PMID 37312287
- Available data/document: Publications: NCT03030274 — http://pubmed.ncbi.nlm.nih.gov/31130524/ — Christina Paitazoglou 1, Ramazan Özdemir, Roman Pfister, Martin W Bergmann, Jozef Bartunek, Teoman Kilic, Alexander Lauten, Alexander Schmeisser, Mehdi Zoghi, Stefan Anker, Horst Sievert, Felix Mahfoud_The AFR-PRELIEVE trial: a prospective, non-randomised, pilot study to assess the Atrial Flow Regulator (AFR) in heart failure patients with either preserved or reduced ejection fraction
- Available data/document: Publications: NCT03030274 — http://pubmed.ncbi.nlm.nih.gov/33555114/ — Christina Paitazoglou 1, Martin W Bergmann 1, Ramazan Özdemir 2, Roman Pfister 3, Jozef Bartunek 4, Teoman Kilic 5, Alexander Lauten 6, Alexander Schmeisser 7, Mehdi Zoghi 8, Stefan D Anker 6, Horst Sievert 9, Felix Mahfoud 10, AFR-PRELIEVE Investigators_One-year results of the first-in-man study investigating the Atrial Flow Regulator for left atrial shunting in symptomatic heart failure patients: the PRELIEVE study
- Available data/document: Publiactions: NCT03030274 — http://pubmed.ncbi.nlm.nih.gov/34763641/ — Nijad Bakhshaliyev 1, Ramazan Ozdemir 1_The impact of atrial flow regulator implantation on hemodynamic parameters in patients with heart failure